CLINICAL TRIAL: NCT04790032
Title: PharmacOdynaMic Effects of Cangrelor in PatiEnts wIth Acute or chronIc Coronary Syndrome Undergoing Percutaneous Coronary Intervention (POMPEII Registry)
Brief Title: Pharmacodynamic Effects of Cangrelor in ACS or CCS Patients Undergoing PCI (POMPEII Registry)
Acronym: POMPEII
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Giuseppe Gargiulo, Principal investigator, Federico II University
Other Study IDs: POMPEII Registry
Record Dates: First submitted 2021-03-04; First posted 2021-03-10 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Percutaneous Coronary Intervention
Keywords: Cangrelor; Acute coronary syndrome; Chronic coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — cangrelor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Cangrelor — All patients receiving Cangrelor during PCI will be enrolled and analyzed for platelet function tests.

SUMMARY:
This prospective registry was designed to carefully investigate the pharmacodynamic (PD) effects of cangrelor in all patients undergoing percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
There is huge interest in achieving fast and immediate antiplatelet effect at the time of PCI, particularly in acute myocardial infarction and Cangrelor is an intravenous antagonist of the P2Y12 receptor characterized by rapid, potent, predictable, and reversible platelet inhibition. However, there are limited pharmacodynamic data exploring the effects of this drug in the various clinical settings at the approved dosages and with current gold standard methods for testing platelet reactivity. More importantly, there are no data on rates and predictors of high residual platelet reactivity (HRPR) in patients treated with cangrelor. Therefore the present study aims at building up a large prospective registry of pharmacodynamic data obtained by light transmittance aggregometry (LTA), multiplate analysis and verifynow system in patients undergoing PCI and receiving cangrelor.

This study is designed as a single-center prospective registry. Investigators at University Hospital of Naples Federico II will enroll patients, collect blood samples, perform platelet function tests and collect clinical and demographic information.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients undergoing PCI and receiving cangrelor administration will be eligible for inclusion in the study.

Exclusion Criteria:

* only those not providing consent to blood/data collection will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with Acute (ACS) or Chronic coronary syndrome (CCS) undergoing PCI and receiving cangrelor administration.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Inhibition of platelet activity (IPA, %) with LTA-ADP 20 µmol/l | 30 minutes
  Platelet inhibition assessed with LTA-ADP 20 µmol/l at 30 minutes and after infusion stop

SECONDARY OUTCOMES:
Maximum platelet aggregation (MPA) with LTA-ADP 20 µmol/l | 30 minutes
  Platelet aggregation assessed with LTA-ADP 20 µmol/l at 30 minutes and after infusion stop
Rates of High Residual Platelet Reactivity (HRPR) with LTA-ADP 20 µmol/l defined as MPA>59% | 30 minutes
  High platelet aggregation assessed with LTA-ADP 20 µmol/l at 30 minutes and after infusion stop
Inhibition of platelet activity (IPA, %) with LTA-ADP 5 µmol/l | 30 minutes
  Platelet inhibition assessed with LTA-ADP 5 µmol/l at 30 minutes and after infusion stop
Maximum platelet aggregation (MPA) with LTA-ADP 5 µmol/l | 30 minutes
  Platelet aggregation assessed with LTA-ADP 5 µmol/l at 30 minutes and after infusion stop
Rates of High Residual Platelet Reactivity with LTA-ADP 5 µmol/l defined as MPA>46% | 30 minutes
  High platelet aggregation assessed with LTA-ADP 5 µmol/l at 30 minutes and after infusion stop
Area under the curve (AUC) at Multiplate with ADP test | 30 minutes
  Platelet aggregation assessed with Multiplate ADP test at 30 minutes and after infusion stop
Rates of HRPR defined as Multiplate AUC >46 U | 30 minutes
  High platelet aggregation assessed with Multiplate ADP test at 30 minutes and after infusion stop
P2Y12 Reaction Unit (PRU) at VerifyNow | 30 minutes
  Platelet aggregation assessed with VerifyNow ADP test at 30 minutes and after infusion stop
Rates of HRPR defined as VerifyNow PRU >208 | 30 minutes
  High platelet aggregation assessed with VerifyNow ADP test at 30 minutes and after infusion stop
Platelet aggregation, inhibition and HRPR by LTA, Multiplate and VerifyNow | After stop of cangrelor infusion
  Platelet aggregation, inhibition and HRPR by LTA, Multiplate and VerifyNow few hours after cangrelor infusion interruption
Clinical outcomes at 30 days | 30 day
  Ischemic and bleeding outcomes at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Gargiulo, MD, PhD, Principal Investigator — Department of Advanced Biomedical Sciences, University Federico II of Naples, Italy; Giovanni Esposito, MD, PhD, Study Chair — Department of Advanced Biomedical Sciences, University Federico II of Naples, Italy
Locations (1):
- University Federico II of Naples, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gargiulo G, Esposito G, Avvedimento M, Nagler M, Minuz P, Campo G, Gragnano F, Manavifar N, Piccolo R, Tebaldi M, Cirillo P, Hunziker L, Vranckx P, Leonardi S, Heg D, Windecker S, Valgimigli M. Cangrelor, Tirofiban, and Chewed or Standard Prasugrel Regimens in Patients With ST-Segment-Elevation Myocardial Infarction: Primary Results of the FABOLUS-FASTER Trial. Circulation. 2020 Aug 4;142(5):441-454. doi: 10.1161/CIRCULATIONAHA.120.046928. Epub 2020 Jun 27. PMID 32795098
- [Background] Sibbing D, Aradi D, Alexopoulos D, Ten Berg J, Bhatt DL, Bonello L, Collet JP, Cuisset T, Franchi F, Gross L, Gurbel P, Jeong YH, Mehran R, Moliterno DJ, Neumann FJ, Pereira NL, Price MJ, Sabatine MS, So DYF, Stone GW, Storey RF, Tantry U, Trenk D, Valgimigli M, Waksman R, Angiolillo DJ. Updated Expert Consensus Statement on Platelet Function and Genetic Testing for Guiding P2Y12 Receptor Inhibitor Treatment in Percutaneous Coronary Intervention. JACC Cardiovasc Interv. 2019 Aug 26;12(16):1521-1537. doi: 10.1016/j.jcin.2019.03.034. Epub 2019 Jun 12. PMID 31202949
- [Background] Angiolillo DJ, Rollini F, Storey RF, Bhatt DL, James S, Schneider DJ, Sibbing D, So DYF, Trenk D, Alexopoulos D, Gurbel PA, Hochholzer W, De Luca L, Bonello L, Aradi D, Cuisset T, Tantry US, Wang TY, Valgimigli M, Waksman R, Mehran R, Montalescot G, Franchi F, Price MJ. International Expert Consensus on Switching Platelet P2Y12 Receptor-Inhibiting Therapies. Circulation. 2017 Nov 14;136(20):1955-1975. doi: 10.1161/CIRCULATIONAHA.117.031164. Epub 2017 Oct 30. PMID 29084738
- [Result] Gargiulo G, Cirillo P, Sperandeo L, Castiello DS, Manzi L, Forzano I, Florimonte D, Simonetti F, Canonico ME, Avvedimento M, Paolillo R, Spinelli A, Buongiorno F, Serafino LD, Spaccarotella CAM, Franzone A, Piccolo R, Stabile E, Valgimigli M, Esposito G. Pharmacodynamic effects of cangrelor in patients with acute or chronic coronary syndrome undergoing percutaneous coronary intervention: the POMPEII Registry. EuroIntervention. 2025 May 16;21(10):560-570. doi: 10.4244/EIJ-D-24-00757. PMID 40375762